CLINICAL TRIAL: NCT01703377
Title: Effect of Constraining Joint Motions on Postural Control
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201203044RIC
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Healthy Adults

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A major advantage of understanding a neural control scheme is able to simultaneously perform multiple tasks based on the Uncontrolled Manifold (UCM) hypothesis by taking advantage of motor redundancy. The present study aims to investigate this hypothesis further by examining the effect of artificially eliminating knee and lumbar-thoracic joint motions on postural control when the arms performing targeting task simultaneously in standing. Subjects (Younger group: 20~35 years old; Elder group: 60~85 years old) will execute a targeting task with and without an additional ball-balancing task in standing with free joint motions and with restricted joint motions. The investigators expect to recruit 50 subjects for each group. Analyses of joint configuration variance on the stability of the center of mass (COM) position and the hand path will be performed using the UCM method of variance analysis. This method partitions joint configuration variance into one component consistent with the use of motor abundance and a component that leads to COM position or hand path variability. Furthermore, the differences between the younger group and the elder group will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Participants are healthy with no self-reported neurological deficits, musculoskeletal conditions or motion sickness that affected their ability to maintain stable upright posture.

Exclusion Criteria:

Participants are healthy with self-reported neurological deficits, musculoskeletal conditions or motion sickness that affected their ability to maintain stable upright posture.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults from 18-65 years old
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-04; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Hsu, PhD, Principal Investigator — National Taiwan University
Locations (1):
- School & Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University, Taipei, Taiwan